CLINICAL TRIAL: NCT05572203
Title: Deep Nutritional Phenotyping of Adult Crohn's Disease Patients: a Focus on Protein Intake and Sarcopenia
Brief Title: Phenotyping of Adult Crohn's Focusing on Sarcopenia
Acronym: PACS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 21044; 287471 (Other: The Integrated Research Application System (IRAS))
Record Dates: First submitted 2022-07-26; First posted 2022-10-07 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Inflammatory Bowel Diseases; Sarcopenia; Digestive System Disease; Nutrition, Healthy; Protein Malabsorption; Crohn Disease
Keywords: Labelled protein; protein; muscle protein synthesis; muscle mass; sarcopenia; Inflammatory bowel disease; Crohn's disease; nutrition; DEXA; 13C/2H-labelled amino acids
MeSH Terms: conditions — Inflammatory Bowel Diseases; Sarcopenia; Digestive System Diseases; Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy group (Control group ) (Active Comparator): This group will include healthy participants matching Crohn's group
  Interventions: Dietary Supplement: Intrinsically labelled protein
- Crohn's group or patients group (Experimental): This group will include patients with Crohn's disease.
  Interventions: Dietary Supplement: Intrinsically labelled protein

INTERVENTIONS:
Dietary Supplement: Intrinsically labelled protein — It is a protein drink that includes Intrinsically labelled Casein ( from Arla Foods), 13C/2H-labelled Spirulina (from CK Isotopes), and 13C/2H-labelled amino acids (from CK Isotopes)
  Other Names: Intrinsically labelled Casein

SUMMARY:
Inflammatory bowel disease (IBD) includes two idiopathic chronic relapsing and remitting inflammatory conditions affecting the gastrointestinal (GI) tract: Crohn's disease (CD) and ulcerative colitis (UC)Malnutrition and significant alteration of body composition are common in inflammatory bowel disease patients, whereby the prevalence of malnutrition may be up to 82.8% in CD patients with active disease, and up to 38.9% in CD patients in remission. Many CD patients have low muscle mass and function (sarcopenia) with drivers of such pathophysiology unknown. 41.6% of CD patients with sarcopenia require surgery, with the surgical trauma and resulting inactivity leading to further muscle mass loss such that the chronic inflammatory insult associated with refractory disease may be linked to advanced muscle mass depletion. The majority of adult CD patients have low muscle mass even in clinical remission indicating the poorly reversible nature of this phenomenon. Chronic disease burden may therefore be important in the accentuation of muscle loss.

Muscle mass is maintained through the daily balance of MPS and muscle protein breakdown (MPB), with the essential amino acid (EAA) components of a meal and muscle contraction being the primary stimulators of MPS. Patients with active CD show a significant decrease in the expression of proteins in hypertrophic signalling pathways (Akt, P70S6K1) with no change in the expression of atrophic signalling (MAFbx, MuRF1). Also, adult CD patients with established disease consume less protein compared to matched healthy volunteers (HV). Furthermore, the intestinal motility, measured using cine-MRI, is reduced in active CD, possibly further decreasing intestinal digestion and absorption of dietary peptides. In general, the malabsorption is a major contributing factor to malnourishment in CD. It has been shown that in male paediatric patients with long-term CD, muscle metabolism is perturbed by a negative branched-chain amino acid balance in the forearm, with this variable linked to lower appendicular muscle mass, higher muscle fatigue and reduced protein intake, CD may have a significant effect on protein digestion and absorption, and blunt the MPS response to feeding, leading to a chronic muscle mass reduction that may persist even when in remission.

The EAA components of a protein meal are crucial for the stimulation of muscle protein synthesis (MPS), and all the EAA/leucine play a key role in driving MPS. Low serum levels EAA/leucine have been reported in CD but their role in the aetiology of sarcopenia in CD is unknown.

Further, how CD affects the protein digestion/absorption and how this contributes to low EAA/leucine unclear. Recent advances in stable isotope tracer techniques using a dual tracer methodology now enable a more accurate determination of protein digestibility. By following the appearance of intrinsically labelled AAs into the blood upon digestion of the intrinsically labelled protein, alongside the appearance of label-free AAs, protein digestibility can be accurately determined. Further, by collecting a muscle biopsy postprandially, the direct incorporation of AA from the digested protein into the muscle can be determined- providing a gold standard method for investigating anabolic resistance.

Project aim is to use an intrinsically labelled casein to investigate protein digestion, absorption and MPS responses in CD patients.

To achieve this, investigators will investigate protein digestion, absorption and muscle protein synthesis responses in Crohn's disease patients and healthy volunteers by utilising intrinsically labelled protein.

ELIGIBILITY:
Inclusion Criteria for Healthy group

1. Aged 18 years or older
2. BMI <30 kg/m2/
3. No previous known bowel disease
4. Be able to provide written informed consent & participate fully in all aspects of the study.

Inclusion Criteria for Crohn's group:

1. Aged 18 years or older.
2. BMI <30 kg/m2
3. Documented diagnosis of CD previously confirmed by endoscopy and histology at least 2 years prior to enrolment.
4. Active CD defined as HBI >4 and CRP >5g/l or FCP >250ug/g or as deemed through endoscopy or cross sectional imaging.
5. Previous biologic or immunosuppressant exposure
6. Previous CD-related intestinal surgery
7. Able to participate fully in all aspects of the study
8. Written informed consent obtained and documented

Exclusion Criteria for Healthy group

1. Aged 18 years or older
2. BMI <30 kg/m2/
3. No previous known bowel disease
4. Be able to provide written informed consent & participate fully in all aspects of the study.

Exclusion Criteria for Crohn's group

1. A current diagnosis of ulcerative colitis, indeterminate colitis, microscopic colitis, or diverticular disease-associated colitis
2. A diagnosis of short-bowel syndrome
3. Use of systemic corticosteroids for CD (2 continuous weeks or more) within 3 months prior to enrolment, or use of any medications for HVs and CD, in the opinion of the investigator, may interfere with the subject's ability to participate fully in the study.
4. Serious underlying disease other than CD that, in the opinion of the investigator, may interfere with the subject's ability to participate fully in the study.
5. History of active alcohol or drug abuse that, in the opinion of the investigator, may interfere with the subject's ability to comply with the study procedures.
6. Pregnancy or breastfeeding.
7. Contraindications for DEXAscanning e.g. x-ray within last 7 days.
8. Allergy to milk, , or casein

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Postprandial muscle protein synthesis. | Change from baseline 4 hours (Two time points)
  Postprandial muscle bound [ring-D5]-Phenylalanine, [5,5,5-D3]-Leucine as measured through mass spectrometry

SECONDARY OUTCOMES:
Appearance/ digestibility of plasma Amino Acid in blood. | blood samples will be taken at regular intervals up to 240 minutes (max 120ml total blood draw post protein drink). 12-time points
  Postprandial plasma [ring-D5]-Phenylalanine, [5,5,5-D3]-Leucine as measured through mass spectrometry
Muscle mRNA expression of anabolic and catabolic | Change from baseline at 4 hours (Two time points).
  The mRNA expression of transcripts involved anabolic and catabolic signalling pathways as measured through RT-qPCR (Applied Biosystems).
Muscle protein expression of anabolic and catabolic pathway. | Change from baseline at 4 hours (Two time points).
  Muscle protein expression of anabolic and catabolic pathway signalling proteins
Serum Cytokines levels of IL-1 | Only at baseline.
  As measured using ELISAs
Serum Cytokines levels of IL-6 | Only at baseline.
  As measured using ELISAs
Serum Cytokines levels of IL-10 | Only at baseline.
  As measured using ELISAs
Serum Cytokines levels of CRP | Only at baseline.
  As measured using ELISAs (IBDQ)
Serum Cytokines levels of TNF | Only at baseline.
  Daily energy intake and dietary macronutrient composition
Appendicular Lean Mass (ALM) to Height Ratio (Kg/Height2) through DEXA scan | Only at baseline
  - It will be assessed via DEXA scan using a GE Lunar Prodigy DEXA scanner housed in the University of Nottingham's David Greenfield unit. The scan will be a whole-body scan for total body composition measurement including ALM to height. The scans will be analysed using the scanners inbuilt Corescan software. Regional measurements will be taken post scan using custom analysis functions within the Corescan software.
Appendicular skeletal muscle index (ASMI; kg/m2) through DEXA scan. | Only at baseline
  It will be assessed via DEXA scan using a GE Lunar Prodigy DEXA scanner housed in the University of Nottingham's David Greenfield unit. The scan will be a whole-body scan for total body composition measurement including ASMI. The scans will be analysed using the scanners inbuilt Corescan software. Regional measurements will be taken post scan using custom analysis functions within the Corescan software
Skeletal muscle index (SMI; kg/m2) through DEXA scan. | Only at baseline
  It will be assessed via DEXA scan using a GE Lunar Prodigy DEXA scanner housed in the University of Nottingham's David Greenfield unit. The scan will be a whole-body scan for total body composition measurement including SMI. The scans will be analysed using the scanners inbuilt Corescan software. Regional measurements will be taken post scan using custom analysis functions within the Corescan software.
Skeletal Muscle Mass Percentage (SMM; %) through DEXA scan. | Only at baseline
  It will be assessed via DEXA scan using a GE Lunar Prodigy DEXA scanner housed in the University of Nottingham's David Greenfield unit. The scans will be analysed using the scanners inbuilt Corescan software. Regional measurements will be taken post scan using custom analysis functions within the Corescan software.
Total Body Fat Percentage (BF; %) through DEXA scan. | Only at baseline
  It will be assessed via DEXA scan using a GE Lunar Prodigy DEXA scanner housed in the University of Nottingham's David Greenfield unit. The scans will be analysed using the scanners inbuilt Corescan software. Regional measurements will be taken post scan using custom analysis functions within the Corescan software.
Fat Mass Index (FMI; kg/m2) through DEXA scan. | Only at baseline
  It will be assessed via DEXA scan using a GE Lunar Prodigy DEXA scanner housed in the University of Nottingham's David Greenfield unit. The scans will be analysed using the scanners inbuilt Corescan software. Regional measurements will be taken post scan using custom analysis functions within the Corescan software.
Resting Metabolic Rate (RMR) through DEXA scan. | Only at baseline
  It will be assessed via DEXA scan using a GE Lunar Prodigy DEXA scanner housed in the University of Nottingham's David Greenfield unit. The scans will be analysed using the scanners inbuilt Corescan software. Regional measurements will be taken post scan using custom analysis functions within the Corescan software.
Muscle Strength through Handgrip | Only at baseline
  Handgrip Dynamometers are instruments for measuring the maximum isometric strength of the hand and forearm muscles
Muscle Strength through Cybex Dynamometer | Only at baseline
  A CYBEX Isokinetic Test is used to measure the maximum strength of a joint throughout its available range-of-motion (ROM).
Daily physical activity | Only at baseline
  Physical activity as measured with IPAQ
Quality of life for Crohn's disease patients | Only at baseline
  measured through the Short Quality of Life Questionnaire for Inflammatory Bowel Disease
Dietary intake of one day before the experiment day. | Only at baseline
  As analysed by using intake24 website; https://intake24.co.uk/info/output . The participant will be received email included the link to fill it by what they intake on this day.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Benjamin J, Makharia GK, Kalaivani M, Joshi YK. Nutritional status of patients with Crohn's disease. Indian J Gastroenterol. 2008 Sep-Oct;27(5):195-200. PMID 19112190
- [Background] Brook MS, Wilkinson DJ, Phillips BE, Perez-Schindler J, Philp A, Smith K, Atherton PJ. Skeletal muscle homeostasis and plasticity in youth and ageing: impact of nutrition and exercise. Acta Physiol (Oxf). 2016 Jan;216(1):15-41. doi: 10.1111/apha.12532. Epub 2015 Jun 21. PMID 26010896
- [Background] Bukhari SS, Phillips BE, Wilkinson DJ, Limb MC, Rankin D, Mitchell WK, Kobayashi H, Greenhaff PL, Smith K, Atherton PJ. Intake of low-dose leucine-rich essential amino acids stimulates muscle anabolism equivalently to bolus whey protein in older women at rest and after exercise. Am J Physiol Endocrinol Metab. 2015 Jun 15;308(12):E1056-65. doi: 10.1152/ajpendo.00481.2014. Epub 2015 Mar 31. PMID 25827594
- [Background] Chiba T, Suzuki K, Matsumoto T. Plasma-Free Amino Acid Profiles in Crohn's Disease: Relationship With the Crohn Disease Activity Index. Clin Med Insights Gastroenterol. 2018 Jul 30;11:1179552218791173. doi: 10.1177/1179552218791173. eCollection 2018. PMID 30083065
- [Background] Cuthbertson D, Smith K, Babraj J, Leese G, Waddell T, Atherton P, Wackerhage H, Taylor PM, Rennie MJ. Anabolic signaling deficits underlie amino acid resistance of wasting, aging muscle. FASEB J. 2005 Mar;19(3):422-4. doi: 10.1096/fj.04-2640fje. Epub 2004 Dec 13. PMID 15596483
- [Background] Dalton M, Blundell J, Finlayson GS. Examination of food reward and energy intake under laboratory and free-living conditions in a trait binge eating subtype of obesity. Front Psychol. 2013 Oct 21;4:757. doi: 10.3389/fpsyg.2013.00757. eCollection 2013. PMID 24155732
- [Background] Davies A, Nixon A, Muhammed R, Tsintzas K, Kirkham S, Stephens FB, Moran GW. Reduced skeletal muscle protein balance in paediatric Crohn's disease. Clin Nutr. 2020 Apr;39(4):1250-1257. doi: 10.1016/j.clnu.2019.05.017. Epub 2019 May 25. PMID 31178247
- [Background] Devi S, Varkey A, Sheshshayee MS, Preston T, Kurpad AV. Measurement of protein digestibility in humans by a dual-tracer method. Am J Clin Nutr. 2018 Jun 1;107(6):984-991. doi: 10.1093/ajcn/nqy062. PMID 29771297
- [Background] Hartman C, Eliakim R, Shamir R. Nutritional status and nutritional therapy in inflammatory bowel diseases. World J Gastroenterol. 2009 Jun 7;15(21):2570-8. doi: 10.3748/wjg.15.2570. PMID 19496185
- [Background] Khalaf A, Nowak A, Menys A, Marciani L, Taylor SA, Spiller RC, Gowland PA, Moran GW, Hoad CL. Cine MRI assessment of motility in the unprepared small bowel in the fasting and fed state: Beyond the breath-hold. Neurogastroenterol Motil. 2019 Jan;31(1):e13466. doi: 10.1111/nmo.13466. Epub 2018 Sep 19. PMID 30230099
- [Background] Li S, Ney M, Eslamparast T, Vandermeer B, Ismond KP, Kroeker K, Halloran B, Raman M, Tandon P. Systematic review of nutrition screening and assessment in inflammatory bowel disease. World J Gastroenterol. 2019 Jul 28;25(28):3823-3837. doi: 10.3748/wjg.v25.i28.3823. PMID 31391776
- [Background] Moshfegh AJ, Rhodes DG, Baer DJ, Murayi T, Clemens JC, Rumpler WV, Paul DR, Sebastian RS, Kuczynski KJ, Ingwersen LA, Staples RC, Cleveland LE. The US Department of Agriculture Automated Multiple-Pass Method reduces bias in the collection of energy intakes. Am J Clin Nutr. 2008 Aug;88(2):324-32. doi: 10.1093/ajcn/88.2.324. PMID 18689367
- [Background] Moughan PJ, Wolfe RR. Determination of Dietary Amino Acid Digestibility in Humans. J Nutr. 2019 Dec 1;149(12):2101-2109. doi: 10.1093/jn/nxz211. PMID 31529051
- [Background] Neurath MF. Cytokines in inflammatory bowel disease. Nat Rev Immunol. 2014 May;14(5):329-42. doi: 10.1038/nri3661. Epub 2014 Apr 22. PMID 24751956
- [Background] Pizzoferrato M, de Sire R, Ingravalle F, Mentella MC, Petito V, Martone AM, Landi F, Miggiano GAD, Mele MC, Lopetuso LR, Schiavoni E, Napolitano D, Turchini L, Poscia A, Nicolotti N, Papa A, Armuzzi A, Scaldaferri F, Gasbarrini A. Characterization of Sarcopenia in an IBD Population Attending an Italian Gastroenterology Tertiary Center. Nutrients. 2019 Sep 24;11(10):2281. doi: 10.3390/nu11102281. PMID 31554166
- [Background] Rocha R, Santana GO, Almeida N, Lyra AC. Analysis of fat and muscle mass in patients with inflammatory bowel disease during remission and active phase. Br J Nutr. 2009 Mar;101(5):676-9. doi: 10.1017/S0007114508032224. PMID 18631418
- [Background] Ryan E, McNicholas D, Creavin B, Kelly ME, Walsh T, Beddy D. Sarcopenia and Inflammatory Bowel Disease: A Systematic Review. Inflamm Bowel Dis. 2019 Jan 1;25(1):67-73. doi: 10.1093/ibd/izy212. PMID 29889230
- [Background] Silverberg MS, Satsangi J, Ahmad T, Arnott ID, Bernstein CN, Brant SR, Caprilli R, Colombel JF, Gasche C, Geboes K, Jewell DP, Karban A, Loftus EV Jr, Pena AS, Riddell RH, Sachar DB, Schreiber S, Steinhart AH, Targan SR, Vermeire S, Warren BF. Toward an integrated clinical, molecular and serological classification of inflammatory bowel disease: report of a Working Party of the 2005 Montreal World Congress of Gastroenterology. Can J Gastroenterol. 2005 Sep;19 Suppl A:5A-36A. doi: 10.1155/2005/269076. PMID 16151544
- [Background] van Langenberg DR, Della Gatta P, Hill B, Zacharewicz E, Gibson PR, Russell AP. Delving into disability in Crohn's disease: dysregulation of molecular pathways may explain skeletal muscle loss in Crohn's disease. J Crohns Colitis. 2014 Jul;8(7):626-34. doi: 10.1016/j.crohns.2013.11.024. Epub 2013 Dec 13. PMID 24332699
- [Background] Wardle RA, Thapaliya G, Nowak A, Radford S, Dalton M, Finlayson G, Moran GW. An Examination of Appetite and Disordered Eating in Active Crohn's Disease. J Crohns Colitis. 2018 Jun 28;12(7):819-825. doi: 10.1093/ecco-jcc/jjy041. PMID 29617753
- [Background] Wolfe RR. Branched-chain amino acids and muscle protein synthesis in humans: myth or reality? J Int Soc Sports Nutr. 2017 Aug 22;14:30. doi: 10.1186/s12970-017-0184-9. eCollection 2017. PMID 28852372